CLINICAL TRIAL: NCT06947291
Title: A Multicenter, Open-label, Phase II Clinical Study to Evaluate the Safety and Efficacy of Glumetinib Combined With Docetaxel for Injection (Albumin-bound) in Patients With Advanced Gastric Cancer/Gastroesophageal Junction Adenocarcinoma and Other Solid Tumors With MET Overexpression and/or Amplification
Brief Title: Safety and Efficacy of Glumetinib Combined With Docetaxel for Injection (Albumin-bound) in Patients With Advanced Gastric Cancer/Gastroesophageal Junction Adenocarcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYH2065-004
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced Gastric Cancer/Gastroesophageal Junction Adenocarcinoma and Other Solid Tumors
MeSH Terms: interventions — glumetinib; Docetaxel; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Glumetinib combined with Docetaxel for Injection (Albumin-bound) (Experimental): Patients will be administered glumetinib once daily and Docetaxel for Injection (Albumin-bound) by intravenous injection in each 21-day treatment cycle. The treatment will continue until PD, death, intolerable toxicity, or withdrawal at the patient's discretion (whichever occurs first).
  Interventions: Drug: Glumetinib Tablets; Drug: Docetaxel for Injection (Albumin-bound)
- Glumetinib (Active Comparator): Patients will be administered glumetinib once daily in each 21-day treatment cycle. The treatment will continue until PD, death, intolerable toxicity, or withdrawal at the patient's discretion (whichever occurs first).
  Interventions: Drug: Glumetinib Tablets

INTERVENTIONS:
Drug: Glumetinib Tablets — glumetinib once daily once daily under fasting conditions in each 21-day treatment cycle.
Drug: Docetaxel for Injection (Albumin-bound) — Docetaxel for Injection (Albumin-bound) by intravenous injection in each 21-day treatment cycle.
  Arms: Glumetinib combined with Docetaxel for Injection (Albumin-bound)

SUMMARY:
The trial consists of Stage 1 (including dose escalation and dose expansion) and Stage 2 (proof-of-concept study). Among them, Stage 2 adopts a randomized, controlled, open-label, and multicenter design.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients who are able to understand and voluntarily sign the written ICF;
* 2. Male or female patients aged ≥ 18 years (inclusive);
* 3. Patients with advanced solid tumors diagnosed by pathology or cytology;
* 4. Patients with a past medical history showing either negative or positive Her-2 expression can be enrolled. For those with unknown Her-2 expression, the Her-2 status needs to be determined before enrollment. For patients with positive Her-2 expression, their previous treatments should include anti-Her-2 drug therapy.
* 5. Overexpression and/or amplification of MET in tumor tissue specimens/blood samples confirmed by the central laboratory.
* 6. There are measurable lesions or non-measurable but evaluable lesions according to RECIST v1.1.
* 7. The Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score is 0 or 1.
* 8. The expected survival time is ≥ 3 months.
* 9. The functions of major organs and bone marrow meet the criteria.

Exclusion Criteria:

* 1. Patients with prior treatment with targeted MET drugs;
* 2. Previous treatments included docetaxel;
* 3. Patients with meningeal metastases, spinal cord compression, symptomatic or progressive brain metastases are not eligible for enrollment.
* 4. Known hypersensitivity or intolerable conditions to any component of the drugs in the study protocol or their excipients.
* 5. According to NCI-CTCAE 5.0, adverse events caused by previous anti-tumor treatment have not recovered to ≤ Grade 1 (excluding toxicities such as Grade 2 alopecia which are judged by the investigator to pose no safety risk).
* 6. Any severe and/or uncontrolled co-existing diseases that may prevent the patient from participating in the study.
* 7. Female patients who are lactating or pregnant; Women of childbearing potential with a positive blood pregnancy test result within 7 days before trial enrollment. Lactating women can participate in this study if they stop breastfeeding, but they must not resume breastfeeding during and after the completion of the study treatment.
* 8. Any male or female patient of childbearing potential who refuses to use a highly effective contraceptive method throughout the trial period and within 6 months after the last administration.
* 9. Those who are unwilling or unable to comply with the study procedures and requirements, or those who, in the judgment of the investigator, are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Dose escalation and cohort expansion phase: The occurrence and frequency of DLT (Dose-Limiting Toxicity) | Up to approximately 24 months after the first patient is enrolled
Dose escalation and cohort expansion phase: the occurrence and frequency of AE (Adverse Events) and SAE (Serious Adverse Events) (in accordance with NCI-CTCAE 5.0) | Up to approximately 24 months after the first patient is enrolled
Dose escalation and cohort expansion phase: Recommended Phase 2 Dose (RP2D) for the combination therapy. | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept phase: Objective Response Rate (ORR) evaluated by the Independent Review Committee (IRC) according to the RECIST 1.1 criteria. | Up to approximately 24 months after the first patient is enrolled

SECONDARY OUTCOMES:
Dose escalation and cohort expansion phase: Evaluated by the Investigator according to the RECIST 1.1 criteria: Objective Response Rate (ORR) | Up to approximately 24 months after the first patient is enrolled
Dose escalation and cohort expansion phase: Evaluated by the Investigator according to the RECIST 1.1 criteria: Disease Control Rate (DCR) | Up to approximately 24 months after the first patient is enrolled
Dose escalation and cohort expansion phase: Evaluated by the Investigator according to the RECIST 1.1 criteria: Duration of Response (DoR) | Up to approximately 24 months after the first patient is enrolled
Dose escalation and cohort expansion phase: Evaluated by the Investigator according to the RECIST 1.1 criteria: Progression-Free Survival (PFS) | Up to approximately 24 months after the first patient is enrolled
Dose escalation and cohort expansion phase: Overall Survival (OS) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study：Evaluated by the Independent Review Committee (IRC) according to the RECIST 1.1 criteria: Disease Control Rate (DCR) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study：Evaluated by the Independent Review Committee (IRC) according to the RECIST 1.1 criteria:Duration of Response (DoR) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study：Evaluated by the Independent Review Committee (IRC) according to the RECIST 1.1 criteria: Progression-Free Survival (PFS) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study： Evaluated by the Investigator according to the RECIST 1.1 criteria: Objective Response Rate (ORR) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study：Evaluated by the Investigator according to the RECIST 1.1 criteria: Disease Control Rate (DCR) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study：Evaluated by the Investigator according to the RECIST 1.1 criteria: Duration of Response (DoR) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study： Evaluated by the Investigator according to the RECIST 1.1 criteria: Progression-Free Survival (PFS) | Up to approximately 24 months after the first patient is enrolled
Proof-of-concept study： Overall Survival (OS) | Up to approximately 24 months after the first patient is enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China